CLINICAL TRIAL: NCT01933230
Title: Trial of Cooling for Patients With Excel Cryo Cooling System in Intracerebral Hemorrhage (ICH)
Acronym: CCSICH
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed due to issues encountered with meeting enrollment goals at our site.
Sponsor: The Cleveland Clinic (Other)
Collaborators: Cryothermic Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13-121-CCSICH
Record Dates: First submitted 2013-08-23; First posted 2013-09-02 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2015-02

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Excel Cryo Cooling System Collar (Other): An Excel Cryo Cooling System collar will be placed around the neck for a 2 hour neck cooling period. This will cool the blood in the neck that goes to the brain causing the brain to become cool. The collar is a standard neck collar used for patients after neck surgery with a modification that allows for the placement of a cooling pack in the collar. The cooling pack is similar to the cooling packs used for sports injuries. The cooling packs will be changed every 20 minutes for the two-hour duration. During the study and for two hours after, we will collect data concerning the brain temperature, body temperature, brain oxygen level and pressure both in the head and in the blood.
  Interventions: Device: Excel Cryo Cooling System

INTERVENTIONS:
Device: Excel Cryo Cooling System — An Excel Cryo Cooling System collar will be place around the neck for two hours. This will cool the blood in the neck that goes to the brain causing the brain to become cool. The collar is a standard neck collar used for patients after neck surgery with a modification that allows for the placement of a cooling pack in the collar. The cooling pack is similar to the cooling packs used for sports injuries. The cooling packs will be changed every 20 minutes for the two-hour duration. During the study and for two hours after, we will collect data concerning the brain temperature, body temperature, brain oxygen level, and pressure both in the head and in the blood.
  2 hour neck cooling period

SUMMARY:
The purpose of this study is to determine if cooling the neck of patients with ICH decreases brain temperature. In addition, the investigators will determine if the device improves the delivery of oxygen to the brain. A third goal is to determine if cooling the neck lowers intracranial pressure (which is often times high in patients after ICH).

DETAILED DESCRIPTION:
This is a non-randomized device efficacy trial. Patients with >20cc Supratentorial ICH and an invasive brain temperature monitor (either Licox or Temperature sensing intracranial pressure device) will be enrolled after consent. The Excel Cryo Cooling System collar will be placed around neck in up to 20 patients for two hours. The goal is to determine the effectiveness of this device in cooling the brain. The collar is a standard neck collar used for patients after neck surgery with a modification that allows for the placement of a cooling pack in the collar that delivers the cold. During the study and for two hours after, the investigators will collect data concerning the brain temperature, body temperature, brain oxygen level and pressure both in the head and in the blood (blood pressure). The investigators will also collect demographic information about you (i.e. age, gender, medical risk factors) and information regarding your current disease process.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with brain injury in the Neurological ICU.
2. Consent from the patient or surrogate decision maker.
3. Warfarin induced intracerebral hemorrhages only after correction of INR to <1.4.

Exclusion Criteria:

1. Cerebellar hemorrhages.
2. Moribund state where the physician team doesn't believe the patient will survive.
3. Patients who are being cared for with the intent of making them comfortable. DNR-CC (by Ohio law).
4. Known history of a blood dyscrasia such as CLL or essential thrombocytosis that could affect inflammation.
5. Known significant carotid artery stenosis (known >50% stenosis by history or incidental hospital imaging). This will not be specifically tested. Patients found to have significant stenosis later in the hospital stay will have their data interpreted separately as well as in the total group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Javier Provencio, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Excel Cryo Cooling System Collar: We will place an Excel Cryo Cooling System collar around your neck for a 2 hour neck cooling period. This will cool the blood in the neck that goes to the brain causing the brain to become cool as well. The collar is a standard neck collar used for patients after neck surgery with a modification that allows for the placement of a cooling pack in the collar that delivers the cold. The cooling pack is similar to, but not the same as, the cooling packs used for sports injuries. The cooling packs will be changed every 20 minutes for the two-hour duration of the study. During the study and for two hours after, we will collect data concerning the brain temperature (if applicable), body temperature, brain oxygen level (if applicable) and pressure both in the head (if applicable) and in the blood (blood pressure).
  Excel Cryo Cooling System: We will place an Excel Cryo Cooling System collar around your neck for two hours.
Period: Overall Study
Arm/Group | Excel Cryo Cooling System Collar
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Excel Cryo Cooling System Collar: We will place an Excel Cryo Cooling System collar around your neck for a 2 hour neck cooling period. The cooling packs will be changed every 20 minutes for the two-hour duration of the study. During the study and for two hours after, we will collect data concerning the brain temperature (if applicable), body temperature, brain oxygen level (if applicable) and pressure both in the head (if applicable) and in the blood (blood pressure).
  We will place an Excel Cryo Cooling System collar around your neck for two hours. The cooling packs will be changed every 20 minutes for the two-hour duration of the study. During the study and for two hours after, we will collect data concerning the brain temperature (if applicable), body temperature, brain oxygen level (if applicable) and pressure both in the head (if applicable) and in the blood (blood pressure).
  2 hour neck cooling period
Arm/Group | Excel Cryo Cooling System Collar
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (2.83)
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2
temperature [Mean (Standard Deviation); unit: degrees celsius] | 37.05 (0.354)

OUTCOME MEASURES:

1. Primary Outcome: Temperature Reduction by 1 Degree Per Hour in the ICU Setting.
Description: Temperature reduction by 1 degree per hour in the Intensive Care Unit setting.
Time Frame: During the 2 hours of neck cooling
Measure: Mean (Standard Deviation); unit: degrees celsius
Groups:
- Excel Cryo Cooling System Collar: We will place an Excel Cryo Cooling System collar around your neck for a 2 hour neck cooling period. This will cool the blood in the neck that goes to the brain causing the brain to become cool as well. The collar is a standard neck collar used for patients after neck surgery with a modification that allows for the placement of a cooling pack in the collar that delivers the cold. The cooling pack is similar to, but not the same as, the cooling packs used for sports injuries. The cooling packs will be changed every 20 minutes for the two-hour duration of the study. During the study and for two hours after, we will collect data concerning the brain temperature (if applicable), body temperature, brain oxygen level (if applicable) and pressure both in the head (if applicable) and in the blood (blood pressure).
Arm/Group | Excel Cryo Cooling System Collar
Number analyzed (Participants) | 2
degrees celsius | 37.05 (0.354)

2. Primary Outcome: To Determine if Neck Cooling Affects Intracranial Pressure
Time Frame: During 2 hours of neck cooling
Reporting Status: Not Posted

3. Primary Outcome: To Determine if Neck Cooling Affects Brain Temperature.
Time Frame: During the 2 hours of neck cooling
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Excel Cryo Cooling System Collar: We will place an Excel Cryo Cooling System collar around your neck for two hours. This will cool the blood in the neck that goes to the brain causing the brain to become cool as well. The collar is a standard neck collar used for patients after neck surgery with a modification that allows for the placement of a cooling pack in the collar that delivers the cold. The cooling pack is similar to, but not the same as, the cooling packs used for sports injuries. The cooling packs will be changed every 20 minutes for the two-hour duration of the study. During the study and for two hours after, we will collect data concerning the brain temperature (if applicable), body temperature, brain oxygen level (if applicable) and pressure both in the head (if applicable) and in the blood (blood pressure).
  2 hour neck cooling period
Arm/Group | Excel Cryo Cooling System Collar
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No